CLINICAL TRIAL: NCT02695524
Title: Effect of Scapula-focused Treatment With Additional Motor Control Exercises on Pain and Disability in Patients With Subacromial Pain Syndrome: A Randomized Controlled Trial
Brief Title: Exercise Application in the Treatment of Patients With Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Anamaria Siriani de Oliveira, Associate Professor, Department of Biomechanics, Medicine and Rehabilitation of Locomotive Apparatus, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1179-1921
Record Dates: First submitted 2016-02-19; First posted 2016-03-01 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Rehabilitation; Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scapula-focused exercises (Active Comparator): Side lying external rotation, prone horizontal abduction , Scapular punch, Knee Push, Full can, D1 Diagonal, three times a week, 8 weeks, 3x10 repetitions
  Interventions: Other: Scapula-focused exercises
- Motor control exercises (Experimental): Towel slide, Scapular Clock, PNF scapular, Inferior Glide modified, Scapular Orientation Exercise, protraction and retraction of scapula, three times a week, 8 weeks, 3x10 repetitions
  Interventions: Other: Scapula-focused exercises; Other: Motor control exercises

INTERVENTIONS:
Other: Scapula-focused exercises
Other: Motor control exercises
  Arms: Motor control exercises

SUMMARY:
This study evaluate the effectiveness of adding neuromuscular exercises with tactile, visual and auditory feedback to a scapula-focused treatment, both emphasizing the periscapular muscles on improvement of disability in patients with subacromial pain syndrome compared to patients receiving only strengthening exercise protocol.

DETAILED DESCRIPTION:
Evidence of the effectiveness conservative treatments in shoulder impingement are in favor the application of specific exercises for scapulothoracic muscles and rotator cuff on pain reduction and improvement of upper limb function, supervised or performed at home, and these same exercises associated with other therapies promote a greater reduction in pain and improvement in disability.

Currently, the evidence of better methodological quality present in the literature13 points out that the performance of motor control exercises focused on the scapula associated with mobilization and stretching generate pain improvement and clinically relevant improvement of the function. The few studies in this area have great methodological diversity with significant limitations. The hypothesis is that patients with subacromial pain syndrome who will receive traditional exercise protocol with the addition of neuromuscular training will show less functional disability, a greater reduction in pain intensity, increase muscle strength and range of motion when compared to the patient group that will receive only the protocol without neuromuscular training, immediately after the intervention, four and eight weeks and four months after randomization and that these benefits are clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial pain syndrome with confirmed positivity in at least three of the five specific orthopedic impact tests: Neer test, Hawkins- Kennedy test, painful arc, external rotation resistance and empty can. Present history of pain in the shoulder lasting more than a week located in the proximal area of the shoulder

Exclusion Criteria:

* Subjects with a history of trauma or shoulder surgery, total rupture of the rotator cuff tendon and biceps, physically active involving the upper limbs or considered active accordance with the short version International Physical Activity Questionnaire (IPAQ). Subjects who have neurological diseases, referred pain in arms (indicative of involvement in the cervical or thoracic region), systemic disease involving the joints such as rheumatoid arthritis or fibromyalgia, the presence of disorders in the wrist such as carpal tunnel syndrome, and have done physical therapy in the shoulder the last six months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gisele H Hotta, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto Medical School, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Publication of data in the form of article:12/2018

REFERENCES:
- [Background] Ludewig PM, Borstad JD. Effects of a home exercise programme on shoulder pain and functional status in construction workers. Occup Environ Med. 2003 Nov;60(11):841-9. doi: 10.1136/oem.60.11.841. PMID 14573714
- [Background] Lombardi I Jr, Magri AG, Fleury AM, Da Silva AC, Natour J. Progressive resistance training in patients with shoulder impingement syndrome: a randomized controlled trial. Arthritis Rheum. 2008 May 15;59(5):615-22. doi: 10.1002/art.23576. PMID 18438933
- [Background] Maenhout AG, Mahieu NN, De Muynck M, De Wilde LF, Cools AM. Does adding heavy load eccentric training to rehabilitation of patients with unilateral subacromial impingement result in better outcome? A randomized, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1158-67. doi: 10.1007/s00167-012-2012-8. Epub 2012 May 12. PMID 22581193
- [Background] Abdulla SY, Southerst D, Cote P, Shearer HM, Sutton D, Randhawa K, Varatharajan S, Wong JJ, Yu H, Marchand AA, Chrobak K, Woitzik E, Shergill Y, Ferguson B, Stupar M, Nordin M, Jacobs C, Mior S, Carroll LJ, van der Velde G, Taylor-Vaisey A. Is exercise effective for the management of subacromial impingement syndrome and other soft tissue injuries of the shoulder? A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Man Ther. 2015 Oct;20(5):646-56. doi: 10.1016/j.math.2015.03.013. Epub 2015 Apr 1. PMID 25920340
- [Background] Michener LA, Walsworth MK, Doukas WC, Murphy KP. Reliability and diagnostic accuracy of 5 physical examination tests and combination of tests for subacromial impingement. Arch Phys Med Rehabil. 2009 Nov;90(11):1898-903. doi: 10.1016/j.apmr.2009.05.015. PMID 19887215
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] de Souza FS, Marinho Cda S, Siqueira FB, Maher CG, Costa LO. Psychometric testing confirms that the Brazilian-Portuguese adaptations, the original versions of the Fear-Avoidance Beliefs Questionnaire, and the Tampa Scale of Kinesiophobia have similar measurement properties. Spine (Phila Pa 1976). 2008 Apr 20;33(9):1028-33. doi: 10.1097/BRS.0b013e31816c8329. PMID 18427325
- [Background] De Mey K, Danneels LA, Cagnie B, Huyghe L, Seyns E, Cools AM. Conscious correction of scapular orientation in overhead athletes performing selected shoulder rehabilitation exercises: the effect on trapezius muscle activation measured by surface electromyography. J Orthop Sports Phys Ther. 2013 Jan;43(1):3-10. doi: 10.2519/jospt.2013.4283. Epub 2012 Nov 16. PMID 23160271
- [Background] Mullaney MJ, McHugh MP, Johnson CP, Tyler TF. Reliability of shoulder range of motion comparing a goniometer to a digital level. Physiother Theory Pract. 2010 Jul;26(5):327-33. doi: 10.3109/09593980903094230. PMID 20557263
- [Background] De Mey K, Danneels L, Cagnie B, Cools AM. Scapular muscle rehabilitation exercises in overhead athletes with impingement symptoms: effect of a 6-week training program on muscle recruitment and functional outcome. Am J Sports Med. 2012 Aug;40(8):1906-15. doi: 10.1177/0363546512453297. Epub 2012 Jul 11. PMID 22785606
- [Background] Reinold MM, Escamilla RF, Wilk KE. Current concepts in the scientific and clinical rationale behind exercises for glenohumeral and scapulothoracic musculature. J Orthop Sports Phys Ther. 2009 Feb;39(2):105-17. doi: 10.2519/jospt.2009.2835. PMID 19194023
- [Background] Kibler WB, Sciascia AD, Uhl TL, Tambay N, Cunningham T. Electromyographic analysis of specific exercises for scapular control in early phases of shoulder rehabilitation. Am J Sports Med. 2008 Sep;36(9):1789-98. doi: 10.1177/0363546508316281. Epub 2008 May 9. PMID 18469224
- [Result] Moezy A, Sepehrifar S, Solaymani Dodaran M. The effects of scapular stabilization based exercise therapy on pain, posture, flexibility and shoulder mobility in patients with shoulder impingement syndrome: a controlled randomized clinical trial. Med J Islam Repub Iran. 2014 Aug 27;28:87. eCollection 2014. PMID 25664288
- [Result] Struyf F, Nijs J, Mollekens S, Jeurissen I, Truijen S, Mottram S, Meeusen R. Scapular-focused treatment in patients with shoulder impingement syndrome: a randomized clinical trial. Clin Rheumatol. 2013 Jan;32(1):73-85. doi: 10.1007/s10067-012-2093-2. Epub 2012 Oct 2. PMID 23053685
- [Result] Armijo-Olivo S, Warren S, Fuentes J, Magee DJ. Clinical relevance vs. statistical significance: Using neck outcomes in patients with temporomandibular disorders as an example. Man Ther. 2011 Dec;16(6):563-72. doi: 10.1016/j.math.2011.05.006. Epub 2011 Jun 12. PMID 21658987

RESULTS

PARTICIPANT FLOW:
Groups:
- Scapula-focused Exercises: Side lying external rotation, prone horizontal abduction , Scapular punch, Knee Push, Full can, D1 Diagonal, three times a week, 8 weeks, 3x10 repetitions
  Scapula-focused exercises
- Motor Control Exercises: Towel slide, Scapular Clock, PNF scapular, Inferior Glide modified, Scapular Orientation Exercise, protraction and retraction of scapula, three times a week, 8 weeks, 3x10 repetitions
  Scapula-focused exercises
  Motor control exercises
Period: Overall Study
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Started | 30 | 30
Completed | 27 | 27
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scapula-focused Exercises | Motor Control Exercises | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10) | 51 (8) | 49 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 30 | 60
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 30 | 30 | 60
Height (m) [Mean (Standard Deviation); unit: meters] | 1.64 (0.08) | 1.64 (0.07) | 1.64 (0.08)
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (4.4) | 29.4 (4.9) | 28.9 (4.6)
Right hand Dominance [Count of Participants; unit: Participants] | 30 | 28 | 58
Painful shoulder on the dominant side [Count of Participants; unit: Participants] | 14 | 18 | 32
Duration of symptoms (mo) [Mean (Standard Deviation); unit: months] | 28 (15) | 29 (33) | 28.8 (26.6)
Medication for pain [Count of Participants; unit: Participants] | 24 | 27 | 51
Body mass (Kg) [Mean (Standard Deviation); unit: Kilograms] | 77 (13.9) | 79.3 (14.2) | 78.1 (14)

OUTCOME MEASURES:

1. Primary Outcome: Change in Functionality Evaluated With Specific Questionnaire
Description: The Brazilian version of Shoulder Pain and Disability Index ranging 0 to 100 points. Lower scores indicate better functionality
Time Frame: baseline, four and eight weeks and sixteen weeks after randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
units on a scale
  baseline | 63.3 [56.4 to 70.1] | 65.7 [57.8 to 74.5]
  4 weeks | 49.8 [41 to 58.7] | 43.5 [33 to 53.9]
  8 weeks | 37.1 [27.6 to 46.6] | 39.7 [28.4 to 50.9]
  16 weeks | 32.8 [23 to 42.5] | 34.2 [23 to 45.4]

2. Secondary Outcome: Change in Intensity of Pain Evaluated by a Scale
Description: Pain Numerical Rating Scale from 0 to 10. Lower values indicate improvement in pain
Time Frame: baseline, four and eight weeks and sixteen weeks after randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 3.7 [2.3 to 5.1] | 3.9 [2.6 to 5.2]
  4 weeks | 2.7 [1.5 to 4] | 1.5 [0.5 to 2.6]
  8 weeks | 1.8 [0.7 to 3] | 1.3 [0.3 to 2.2]
  16 weeks | 0.5 [-0.09 to 1.1] | 1.2 [0.3 to 2.1]

3. Secondary Outcome: Change in Strength Evaluated by Hand Held Dynamometer and the Measures Provided in Kilogram-force (KgF)
Description: Strength of serratus anterior, trapezius muscles, abduction, adduction, internal and external rotation movements the arm with hand held Dynamometer.
Time Frame: baseline, four and eight weeks and sixteen weeks after randomization
Measure: Mean (95% Confidence Interval); unit: Kilogram-force
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
Kilogram-force
  Shoulder abduction baseline | 6.2 [5 to 7.4] | 5.5 [4.3 to 6.6]
  Shoulder abduction 4 weeks | 7.1 [5.8 to 8.5] | 6.3 [5.1 to 7.6]
  Shoulder abduction 8 weeks | 7.9 [6.6 to 9.2] | 7.1 [5.8 to 8.4]
  Shoulder abduction 16 weeks | 7.8 [6.4 to 9.2] | 7 [5.7 to 8.4]
  Shoulder adduction baseline | 7.8 [6.2 to 9.4] | 7.9 [6.5 to 9.4]
  Shoulder adduction 4 weeks | 8.8 [7 to 10.5] | 9 [7.2 to 10.8]
  Shoulder adduction 8 weeks | 9.2 [7.5 to 10.8] | 9.2 [7.6 to 10.8]
  Shoulder adduction 16 weeks | 8.5 [7 to 9.9] | 9 [7.3 to 10.7]
  Shoulder external rotation baseline | 5.8 [4.8 to 6.8] | 5.7 [4.7 to 6.7]
  Shoulder external rotation 4 weeks | 5.9 [5 to 6.8] | 6.1 [5.1 to 7.2]
  Shoulder external rotation 8 weeks | 6.5 [5.7 to 7.3] | 6.5 [5.5 to 7.5]
  Shoulder external rotation 16 weeks | 6.9 [5.8 to 8] | 6.4 [5.3 to 7.4]
  Shoulder Internal rotation baseline | 8.6 [6.7 to 10.4] | 9.4 [7.7 to 11]
  Shoulder Internal rotation 4 weeks | 9.1 [7.4 to 10.8] | 10.4 [8.3 to 12.4]
  Shoulder Internal rotation 8 weeks | 10.4 [8.8 to 12] | 11.4 [9.2 to 13.6]
  Shoulder Internal rotation 16 weeks | 10.3 [8.7 to 11.9] | 10.7 [8.7 to 12.8]
  Serratus Anterior Baseline | 7.2 [5.6 to 8.8] | 6.8 [5 to 8.5]
  Serratus Anterior 4 weeks | 9.1 [7 to 11.1] | 10 [8 to 12]
  Serratus Anterior 8 weeks | 10.3 [8.4 to 12] | 10.8 [8.7 to 13]
  Serratus Anterior 16 weeks | 11.1 [8.8 to 13.3] | 10.6 [8.4 to 12.9]
  Upper Trapezius Baseline | 8.3 [7 to 10] | 8.8 [7.6 to 10]
  Upper Trapezius 4 weeks | 9.8 [8.3 to 11.5] | 11.1 [9.3 to 12.8]
  Upper Trapezius 8 weeks | 11.1 [9.4 to 12.8] | 12.1 [10.4 to 13.8]
  Upper Trapezius 16 weeks | 11 [9.2 to 12.6] | 11.4 [9.5 to 13.2]
  Middle Trapezius Baseline | 4.4 [3.5 to 5.4] | 3.3 [2.7 to 3.9]
  Middle Trapezius 4 weeks | 4.9 [3.9 to 5.9] | 4.1 [3.6 to 4.7]
  Middle Trapezius 8 weeks | 5.1 [4.3 to 6] | 4.4 [3.8 to 5]
  Middle Trapezius 16 weeks | 5.4 [4.3 to 6.5] | 4.6 [3.7 to 5.5]
  Lower Trapezius baseline | 4.3 [3.4 to 5.3] | 3.1 [2.6 to 3.6]
  Lower Trapezius 4 weeks | 4.6 [3.7 to 5.5] | 4 [3.5 to 4.5]
  Lower Trapezius 8 weeks | 5 [4.2 to 5.9] | 4 [3.5 to 4.7]
  Lower Trapezius 16 weeks | 5 [4 to 6] | 4.1 [3.3 to 5]

4. Secondary Outcome: Perceived Change Evaluated by Numerical Scale
Description: Global Perceived Effect Scale ranging -5 to +5 points. Positive values indicate improvement and negative values indicate worsening of symptoms
Time Frame: four, eight weeks and sixteen weeks of randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
units on a scale
  4 weeks | 2 [1 to 2.9] | 2.8 [2.3 to 3.4]
  8 weeks | 2.9 [2.1 to 3.7] | 3.3 [2.8 to 3.8]
  16 weeks | 3.3 [2.7 to 3.9] | 3.1 [2.3 to 3.8]

5. Secondary Outcome: Change in Kinesiophobia Evaluated With Specific Questionnaire
Description: Tampa Scale of Kinesiophobia ranging 17 to 68 points. High scores indicate high degree kinesiophobia
Time Frame: baseline, four and eight weeks and sixteen weeks after randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
units on a scale
  Kinesiophobia baseline | 42.1 [39.2 to 45] | 42.8 [39.7 to 45.9]
  Kinesiophobia 4 weeks | 39.8 [37 to 42.4] | 40.7 [37.8 to 43.6]
  Kinesiophobia 8 weeks | 40.2 [36.8 to 43.5] | 38.9 [35.5 to 42.3]
  Kinesiophobia 16 weeks | 38.7 [34.2 to 40.7] | 37.5 [34.2 to 40.7]

6. Secondary Outcome: Range of Motion Evaluated by Digital Inclinometer and the Measures Provided in Degrees
Description: abduction, adduction, internal and external rotation of the shoulder
Time Frame: baseline, four and eight weeks and sixteen weeks after randomization
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
degrees
  Shoulder Flexion Baseline | 132.5 [118.8 to 146.1] | 129 [116.2 to 141.7]
  Shoulder Flexion 4 weeks | 140.4 [129 to 151.7] | 148.5 [140.3 to 156.6]
  Shoulder Flexion 8 weeks | 148 [138.6 to 157.4] | 147.8 [138.4 to 157.2]
  Shoulder Flexion 16 weeks | 146.6 [137.4 to 155.9] | 149.9 [141.8 to 158]
  Shoulder Abduction Baseline | 125.3 [111.2 to 139.4] | 120.2 [106.4 to 134]
  Shoulder Abduction 4 weeks | 139 [127.4 to 150.6] | 145.2 [137.1 to 153.4]
  Shoulder Abduction 8 weeks | 147.8 [137.1 to 158.4] | 145.5 [135.1 to 155.9]
  Shoulder Abduction 16 weeks | 143.2 [132.3 to 154.1] | 141.3 [129.9 to 152.7]
  Shoulder External Rotation Baseline | 60.1 [59.9 to 76.2] | 60.9 [51.6 to 70.2]
  Shoulder External Rotation 4 weeks | 66.4 [58 to 74.9] | 66.7 [57.8 to 75.6]
  Shoulder External Rotation 8 weeks | 73.7 [66.6 to 80.8] | 68.3 [60 to 76.6]
  Shoulder External Rotation 16 weeks | 71.4 [65.7 to 80.1] | 70 [61.1 to 78.9]
  Shoulder Internal Rotation Baseline | 49.2 [43.1 to 55.2] | 48.6 [43.1 to 54]
  Shoulder Internal Rotation 4 weeks | 53.9 [47.9 to 59.9] | 53.4 [46.7 to 60.1]
  Shoulder Internal Rotation 8 weeks | 59.2 [54.2 to 64.1] | 54.6 [40.3 to 60]
  Shoulder Internal Rotation 16 weeks | 57.1 [51.3 to 62.9] | 54.8 [49.6 to 60]

7. Secondary Outcome: Satisfaction With Treatment Evaluated With Specific Questionnaire
Description: Medrisk Questionnaire ranging 13 to 80 points. High scores indicate satisfaction with treatment
Time Frame: four, eight weeks and sixteen weeks after randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
units on a scale
  Medrisk 4 weeks | 60.8 [58.9 to 62.8] | 63.1 [61.7 to 64.5]
  Medrisk 8 weeks | 61.3 [59.6 to 63] | 63.6 [62.2 to 64.9]
  Medrisk 16 weeks | 62 [60.5 to 63.5] | 63.8 [62.5 to 65.2]

8. Secondary Outcome: Scapula Position Evaluated by Digital Inclinometer and the Measures Provided in Degrees
Description: upward rotation and tilt of the scapula
Time Frame: baseline, four and eight weeks and sixteen weeks after randomization
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
Number analyzed (Participants) | 30 | 30
degrees
  Upward Rotation 0º Baseline | 5.6 [4.1 to 7] | 7 [4.8 to 9.2]
  Upward Rotation 0º 4 weeks | 5.3 [3.8 to 6.8] | 5.7 [4 to 7.4]
  Upward Rotation 0º 8 weeks | 5 [3.4 to 6.5] | 5.7 [3.9 to 7.4]
  Upward Rotation 0º 16 weeks | 5.1 [3.5 to 6.6] | 6.5 [4.6 to 8.4]
  Upward Rotation 90º baseline | 12.8 [9.2 to 15.9] | 13.6 [10.9 to 16.3]
  Upward Rotation 90º 4 weeks | 13.3 [10.7 to 15.4] | 14.5 [11.8 to 17.1]
  Upward Rotation 90º 8 weeks | 15 [12 to 17.7] | 17.6 [14.6 to 20.7]
  Upward Rotation 90º 16 weeks | 16.8 [13.8 to 20] | 20.6 [18.2 to 23.2]
  Upward Rotation 180º baseline | 30.7 [26.4 to 34.2] | 35.5 [31.6 to 39.6]
  Upward Rotation 180º 4 weeks | 37.3 [32.9 to 40.8] | 39.3 [35.8 to 42.9]
  Upward Rotation 180º 8 weeks | 40.9 [36.9 to 44.9] | 44.3 [40.4 to 48.1]
  Upward Rotation 180º 16 weeks | 39.7 [35.5 to 44] | 44.5 [41.5 to 47.6]
  Anterior Tilt 0º baseline | 18.4 [15.6 to 21] | 19 [17 to 21.1]
  Anterior Tilt 0º 4 weeks | 18.4 [15.6 to 21] | 19 [17 to 21.1]
  Anterior Tilt 0º 8 weeks | 19.7 [17 to 22.1] | 19.4 [17.6 to 21.2]
  Anterior Tilt 0º 16 weeks | 18.7 [15.8 to 21.1] | 19.6 [17.6 to 21.6]
  Anterior Tilt 90º baseline | 15 [12.5 to 18] | 14.2 [11.5 to 16.7]
  Anterior Tilt 90º 4 weeks | 14.6 [12.1 to 17] | 13.6 [11.2 to 15.9]
  Anterior Tilt 90º 8 weeks | 15.1 [11.9 to 17.9] | 12.3 [9.7 to 14.9]
  Anterior Tilt 90º 16 weeks | 13.2 [9.8 to 16.4] | 11.7 [8.7 to 14.6]
  Anterior Tilt 180º baseline | 4.3 [-0.2 to 8.9] | 4.2 [1.3 to 7]
  Anterior Tilt 180º 4 weeks | 2 [-2.7 to 6.2] | 3.2 [-0.03 to 6.7]
  Anterior Tilt 180º 8 weeks | 3.1 [-0.9 to 7] | 0.1 [-3.6 to 3.8]
  Anterior Tilt 180º 16 weeks | 0.6 [-4.7 to 4.7] | 0.7 [-3.2 to 4.7]

ADVERSE EVENTS:
Time Frame: 16 weeks after baseline data collection
Description: All-Cause Mortality
Arm/Group | Scapula-focused Exercises | Motor Control Exercises
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scapula-focused Exercises (N=30) | Motor Control Exercises (N=30)
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The limitation of the present study was that the therapist was not blinded concerning treatment assignment and this study did not assess and exclude individuals with central sensitization and high catastrophizing levels

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT02695524/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02695524/ICF_001.pdf